CLINICAL TRIAL: NCT05236400
Title: A Clinical Trial to Verify the Efficacy and Safety of Electric Phlegm Suction System: Prospective, Multi-center, Randomized, Open-label, Pivotal Study
Brief Title: A Clinical Trial to Verify the Efficacy and Safety of Electric Phlegm Suction System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lmeca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LMECA.A1000.CIP
Record Dates: First submitted 2022-01-11; First posted 2022-02-11 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Other Specified Respiratory Disorders

STUDY DESIGN:
Intervention Model Description: This clinical trial is a multicenter, randomized, parallel design, open-label, confirmatory clinical trial.
  Subjects who sign the clinical trial consent form and satisfy the inclusion/exclusion criteria are enrolled in this trial, and are randomly assigned to a test group and a control group in a 1:1 ratio.
  Airway aspiration is performed through the unmanned electric airway aspiration procedure using the test device (LMECA.A1000), which is the test group, and the manual airway aspiration procedure, which is the control group. Subjects will be evaluated for efficacy and safety on Day 3, Day 7, and Day 14 after application of the clinical trial medical device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- unmanned electric phlegm suction system procedure using an investigational device (LMECA.A1000) (Experimental): After participating in a clinical trial and receiving unmanned electric airway aspiration, the efficacy and safety are checked on Day 3 and on Day 7 and Day 14 of the follow-up period.
  Interventions: Device: unmanned electric phlegm suction system procedure using an investigational device (LMECA.A1000)
- Manual phlegm suction system (Active Comparator): After participating in a clinical trial and applying manual airway aspiration, the efficacy and safety are checked on Day 3 and on Day 7 and Day 14 of the follow-up period.
  Interventions: Procedure: Manual phlegm suction system

INTERVENTIONS:
Device: unmanned electric phlegm suction system procedure using an investigational device (LMECA.A1000) — Subjects who have passed the screening test will receive the test device (LMECA.A1000) within a minimum of 3 days and a maximum of 14 days. Efficacy and safety are checked through bronchoscopy before application for clinical trials and 72 hours after application.
  Arms: unmanned electric phlegm suction system procedure using an investigational device (LMECA.A1000)
Procedure: Manual phlegm suction system — Subjects who have passed the screening test will receive a manual phlegm suction system procedure using a catheter by professional medical staff within a minimum of 3 days and a maximum of 14 days. Efficacy and safety are checked through a bronchoscopy before application to clinical trials and 72 hours after application.
  Arms: Manual phlegm suction system

SUMMARY:
Manual airway aspiration is a task performed by a nurse or caregiver and if the nursing/care work is overloaded, it has the disadvantage that airway aspiration cannot be performed an appropriate number of times according to the needs of the patient. Therefore, an electric phlegm suction system that can compensate for the shortcomings has been developed. The purpose of this clinical trial is to compare and evaluate the efficacy and safety of the test device by applying the unmanned electric phlegm suction system procedure using an investigational device (LMECA.A1000) and the conventional manual airway aspiration procedure to the patients who received mechanical ventilation through the artificial airway in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Those aged ≥19 among the in-patients in the intensive care unit of the study site.
* Patients who have been applied with mechanical ventilation through the artificial airway such as tracheal intubation or tracheotomy and have maintained PaO2/FiO2 values above 100mmHg.
* Patients whose application time of mechanical ventilation does not exceed 36 hours
* Those who are expected to see continued application of mechanical ventilation for at least 72 hours after participating in this study

Exclusion Criteria:

* The subject or a legally acceptable representative refuses to participate in the study
* Those who have become pregnant or are planning to become pregnant during the study period
* Patients who need to maintain their plateau pressure with the mechanical ventilation setting of FiO2 exceeding 80% or exceeding Pplat of 30cmH2O.
* Patients with severely lowered immune function such as advanced hematologic malignancy, bone marrow transplantation failure, agranulocytosis, and absolute neutrophil count (ANC) of <500/mm3
* Those with unstable cardiovascular conditions such as arrhythmia accompanied by hemodynamic instability and severe hypoxemia
* Those who continue to bleed due to hemorrhagic causes, including multiple traumas or thrombocytopenia
* If the patient is scheduled for or had performed a solid organ transportation on the day of study participation, or self-recovered through cardiopulmonary resuscitation (CPR)
* Patients with pulmonary disease accompanied by hemoptysis
* In addition, if the medical staff decides that it is not appropriate to apply the investigational device to the subject or perform bronchoscopy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of airway mucosal damage change on 72 hours after application through bronchoscopy results | 72 hours after application of the investigational device
  Comparative assessment on the damage of the airway mucosa between the test group and the control group through bronchoscopy results

SECONDARY OUTCOMES:
Evaluation of airway mucosal damage | At each time point before the application, 7 days, and 14 days after the application of the investigational device
  Comparison of the difference in the degree of damage to the airway mucosa between the test group and the control group
Incidence of mechanical ventilation-related pneumonia | For 2 weeks from the time of investigational device application
  Difference in the incidence of ventilator-associated pneumonia between the test group and the control group group
Rate of investigational device malfunction | For 2 weeks from the time of application of investigational device
  The incidence of malfunction of the investigational device that has been applied to the test group

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Korea University Ansan Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No